CLINICAL TRIAL: NCT00143884
Title: Adjuvant Cellular Immunotherapy for High-Risk Hematologic Malignancy After Allogeneic Stem Cell Transplantation Using Low Intensity Conditioning
Brief Title: Study of Low Intensity Conditioning and Immunotherapy for High-Risk Cancers of the Blood
Status: Terminated | Phase: Phase 2 | Type: Interventional
Sponsor: University of Michigan Rogel Cancer Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Educational/Counseling/Training
Other Study IDs: UMCC 9979
Record Dates: First submitted 2005-08-31; First posted 2005-09-02 (Estimated); Last update posted 2007-04-23 (Estimated); Status verified 2007-01

CONDITIONS: Leukemia; Lymphoma, Low-Grade; Lymphoma, Non-Hodgkin's; Multiple Myeloma; Myelodysplastic Syndromes
MeSH Terms: conditions — Leukemia; Lymphoma, Non-Hodgkin; Multiple Myeloma; Myelodysplastic Syndromes

INTERVENTIONS:
Procedure: Reduced intensity conditioning
Procedure: Prophylactic donor leukocyte infusions

SUMMARY:
This research project will focus on whether it is safe and effective to rely on donor cells to prevent relapse of leukemia, lymphoma, or other blood cancer after bone marrow stem cell transplant.

DETAILED DESCRIPTION:
This research project will focus on whether it is safe and effective to rely on donor cells to prevent relapse of leukemia, lymphoma, or other blood cancer after bone marrow stem cell transplant (SCT). For many patients with these conditions, a bone marrow transplant can be the only chance for cure. The standard type of bone marrow transplant involves giving very high-doses of chemotherapy and radiation to kill all the cancer cells followed by an infusion of bone marrow stem cells from a relative who is a bone marrow match. After the transplant the patient takes anti-rejection drugs for many months to prevent the donor's immune cells from causing a severe reaction called Graft-versus-Host Disease (GVHD), which can even be fatal. However, for some patients with certain types of high-risk cancer even this intense treatment is not effective and the cancer relapses.

Is has been known for many years that some of the bone marrow cells from the donor can kill cancer cells. Recently, it has been discovered that sometimes patients who relapse after a bone marrow SCT can be cured by giving an infusion of donor white blood cells (called a donor leukocyte infusion or DLI). By giving a DLI BEFORE a relapse happens, hopefully relapse can be prevented.

The high doses of chemotherapy and radiation therapy given prior to a standard bone marrow stem cell transplant can make a patient very sick and also increase the chance of getting severe GVHD. In this research study we are going to rely mainly on the donor cells to kill the cancer cells, and patients will receive dosages of chemotherapy that are lower than the usual dosages. It is thought that this low intensity conditioning will make the transplant safer without risking more relapses, however it is not know whether low intensity conditioning is safer than standard conditioning.

ELIGIBILITY:
Patient Inclusion Criteria:

* One of the following hematological malignancies:

  1. Chronic myelogenous leukemia

     1. Accelerated phase
     2. Blast phase
  2. Acute myelogenous leukemia

     1. First or greater complete remission if high risk features: abnormalities of chromosomes with known poor prognosis 5 or 7.
     2. Relapsed or refractory patients with ≤ 30% blasts
     3. Aged 55 years or older in any disease state beyond first remission if blast percentage is < 30%.
  3. Acute lymphoblastic leukemia

     1. First complete remission if high risk features: t(4;11)
     2. Second complete remission if relapse occurs within the first 12 months of therapy
     3. Third or greater complete remission
     4. Relapsed or refractory patients with ≤ 30% blasts
     5. Aged 55 years or old in second in any disease state beyond first remission if blast percentage is < 30%.
  4. Myelodyplastic syndromes

     1. RAEB or RAEB-t patients, 55 years of age or older
     2. Any hematologic malignancy relapsed following autologous or matched related donor allogeneic stem cell transplant provided at least 90 days has elapsed from most recent transplant
  5. Non-Hodgkin's Lymphoma

     1. 55 years or older, who have failed anthracycline containing regimen and do not have any tumor larger than 5 cm in diameter.
     2. Patients with rapidly progressive disease are ineligible.
  6. Multiple myeloma patients, any age, who meet at least one of the following criteria:

     1. disease refractory to conventional chemotherapy such as VAD, pulse decadron, or alkylating agents, OR
     2. chromosomal abnormality by cytogenetics or FISH probe.
  7. Chronic lymphoblastic leukemia patients

     1. Any age
     2. Advanced disease (Rai stage 3 or 4)
     3. Relapsed following/refractory to alkylating agents or nucleoside analog therapy
     4. NOTE: Patients with bulky disease (lymphadenopathy > 5 cm) or progressive disease NOT eligible.
  8. Mantle cell lymphoma

     1. Any age
     2. Disease stage 3 or 4
     3. Lymphadenopathy must not exceed 5 cm in any dimension
  9. Any eligible disease category, any age, if ineligible for myeloablative conditioning because of organ dysfunction or advanced age (55 years or older). Minimum organ function for patients entered on this protocol defined as:

     1. Cardiac: Ejection fraction at least 30%.
     2. Renal: Creatinine <1.5 times normal for age.
     3. Pulmonary: FEV1 and FVC >60%.
     4. Hepatic: Total bilirubin <2.0 and AST/ALT <3 X institutional normal for age.
     5. Performance (adults): Karnofsky score must be at least 60; for pts. under 16, Lansky score must be at least 60.
  10. Low grade lymphoma (small lymphocytic, follicular small cleaved cell, or follicular mixed small cleaved and large cell) must meet the following criteria:

      1. any age
      2. relapsed or refractory disease provided the disease is NOT rapidly progressive
      3. no lymphoma mass or lymph node exceeds 5 cm in greatest dimension
* Age: no age restriction
* Availability of a 6/6 HLA A, B, and DR identical relative who is willing and able to donate allogeneic stem cells
* No active infection
* Serum creatinine less than 1.5 times normal for age
* Serum bilirubin less than 1.5 times normal for age
* Not pregnant.

Patient Exclusion Criteria:

* HIV positive patients not eligible
* Pregnant

Donor Inclusion Criteria:

* 6/6 HLA match for HLA-A, B, and DR
* Age 3-70 years, good general health
* No contraindication to G-CSF stimulation
* No contraindication to leukapheresis of peripheral blood stem cells
* Good general health

Donor Exclusion Criteria:

* HIV positive or history of HIV risk factors
* Presence of other diseases transmissible by blood that pose unacceptable risk to the study subject.
* Pregnant
* Medical or psychological conditions that would make the donor unlikely to tolerate G-CSF injections or leukapheresis

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30
Dates: Start 2000-03

PRIMARY OUTCOMES:
To conduct a phase I-II trial of prophylactic cellular immunotherapy after allogeneic hematopoietic stem cell therapy using low intensity conditioning for high-risk hematological malignancies

SECONDARY OUTCOMES:
To evaluate both surrogate markers of GVHD (with a cytokine panel) and minimal residual disease and correlate these with clinical outcomes during the above trial

CONTACTS AND LOCATIONS:
Overall Officials: John E. Levine, MS MD, Principal Investigator — The Univeristy of Michigan
Locations (1):
- The University of Michigan, Ann Arbor, Michigan, United States